CLINICAL TRIAL: NCT01692938
Title: Evaluation of the Precision of the Microperimetry Function of the Spectral OCT/SLO
Status: Completed | Type: Observational
Sponsor: Optos, PLC (Industry)
Collaborators: Johns Hopkins University (Other); University of Southern California (Other)
Responsible Party: Sponsor
Other Study IDs: OPT1001
Record Dates: First submitted 2012-09-21; First posted 2012-09-26 (Estimated); Results first posted 2015-11-30 (Estimated); Last update posted 2017-05-10 (Actual); Status verified 2017-04

CONDITIONS: Age-Related Macular Degeneration; Geographic Atrophy; Diabetic Retinopathy; Macular Edema; Retinal Vein Occlusion; Central Serous Retinopathy; Pattern Dystrophy of Macula; Epiretinal Membrane; Macular Hole
MeSH Terms: conditions — Macular Degeneration; Geographic Atrophy; Diabetic Retinopathy; Macular Edema; Retinal Vein Occlusion; Central Serous Chorioretinopathy; Epiretinal Membrane; Retinal Perforations

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- No Retinal Disease
- Retinal Disease

SUMMARY:
To conduct a precision study to assess the microperimetry function of the Spectral OCT/SLO. The study will assess variability across measurements taken by three different operator-device configuration across clinical sites, variability between subjects within a given operator-device configuration, and variability within a subject for a single operator-device configuration.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be 21 years of age or older.
* Subjects recruited to Cohort 1 will have no known retinal disease except for refractive errors (-7.5 D to +7.5 diopters).Subjects who are recruited to Cohort 2 will have one or more of the following retinal pathologies: early and intermediate Age-Related Macular Degeneration, Geographic Atrophy, Diabetic Retinopathy (mild, moderate, severe), Macular Edema secondary to Diabetes, Retinal Vein Occlusion, Central Serous Retinopathy, Pattern Dystrophy, Epiretinal Membrane or Macular Hole.
* Subjects who have signed an informed consent form.
* Subjects who can comply with the protocol.

Exclusion Criteria:

* Subjects younger than 21 years of age.
* Subjects who cannot comply with the protocol.
* Subjects who cannot complete the Simple Test procedures
* Subjects who are not available to be testing 3 times during the day (Morning, Mid - Day, and Afternoon).
* Subjects with visual acuity worse than 20/100 (Best Corrected).
* Subjects with dense media opacities.
* Ocular surgery anticipated on the day of the study visit.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Twenty-four subjects, 12 without retinal disease (Cohort 1) and 12 with retinal disease (Cohort 2) will be recruited. Any subjects that do not comply with or complete the study protocol will be replaced to ensure that a total of 24 subjects complete the protocol. Subjects will be screened and recruited based on the Inclusion/Exclusion criteria outlined within this protocol. Subjects fulfilling the stated criteria and who are willing to comply must sign an informed consent prior form to study participation.
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2012-10; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Quan Nguyen, Principal Investigator — Johns Hopkins University
Locations (3):
- United States (3):
  - Retina Group of Florida, Fort Lauderdale, Florida
  - Johns Hopkins Unversity, Baltimore, Maryland
  - Valley Retina Institute, McAllen, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Dates - 10/5/2012 to 11/5/2012. 3 Ophthalmic Clinics.
Period: Overall Study
Arm/Group | No Retinal Disease | Retinal Disease
Started | 16 | 16
Completed | 12 | 12
Not Completed | 4 | 4
Not completed — Protocol Deviation | 1 | 1
Not completed — Study completed prior to site completion | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | No Retinal Disease | Retinal Disease | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Customized [Number; unit: participants]
  21-35 years | 4 | 3 | 7
  36-50 years | 4 | 3 | 7
  51-64 years | 3 | 3 | 6
  65 years or great | 1 | 3 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 6 | 14
  Male | 4 | 6 | 10

OUTCOME MEASURES:

1. Primary Outcome: Standard Deviation and Mean Test Results of Normal and With Pathology Participants Taken by 3 Different Operator-device Configurations
Description: A precision study was conducted that used 3 devices (each with a different operator). Each device was used to measure 4 normal subjects and 4 subjects with relevant eye pathology, with a total of 24 subject eyes (12 normal, 12 with pathology) measured across all three devices. For each subject, one eye was evaluated using 3 tests with repositioning at the start of each test. Test results were given in decibels which is the unit used in microperimetry testing. Overall mean and standard deviation in decibels were calculated for the two groups: normal and with pathology.
Time Frame: 1 Month
Measure: Mean (Standard Deviation); unit: decibels
Arm/Group | No Retinal Disease | Retinal Disease
Number analyzed (Participants) | 12 | 12
decibels | 16.16 (1.735) | 12.23 (3.508)

2. Primary Outcome: Repeatability of Microperimetry Tests in Normal and With Pathology Participants Based on 3 Microperimetry Tests Taken for Each Participant for a Given Operator-device Combination.
Description: A precision study was conducted that used 3 devices (each with a different operator). Each device was used to measure 4 normal subjects and 4 subjects with relevant eye pathology, with a total of 24 subject eyes (12 normal, 12 with pathology) measured across all three devices. Test results were given in decibels as that is the standard measurement in microperimetry testing. For each subject, one eye was evaluated using 3 microperimetry tests with repositioning at the start of each test. Overall Repeatability SD and Repeatability SD Limit were calculated for the two groups: normal and with pathology.
Time Frame: 1 Month
Measure: Mean (Standard Deviation); unit: decibels
Arm/Group | No Retinal Disease | Retinal Disease
Number analyzed (Participants) | 12 | 12
decibels
  Repeatability SD | 16.16 (0.531) | 12.23 (0.682)
  Repeatability SD Limit | 16.16 (1.49) | 12.23 (1.91)

ADVERSE EVENTS:
Arm/Group | No Retinal Disease | Retinal Disease
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 0/16 | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less